CLINICAL TRIAL: NCT00600873
Title: Pharmacokinetics and Nitrative-Oxidative Stress Pharmacodynamics in Amyotrophic Lateral Sclerosis Subjects Taking Daily High-Dose R(+) Pramipexole Dihydrochloride for Six Months
Brief Title: R(+)PPX High Dose Treatment of ALS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bennett, James P., Jr., M.D., Ph.D. (Individual)
Responsible Party: James P. Bennett Jr. M.D. Ph.D. Sponsor, Virginia Commonwealth University
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 13023
Expanded Access: Available
Record Dates: First submitted 2008-01-05; First posted 2008-01-25 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: neuroprotection; oxidative stress
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): patients with early ALS
  Interventions: Drug: R(+) pramipexole dihydrochloride monohydrate

INTERVENTIONS:
Drug: R(+) pramipexole dihydrochloride monohydrate — 100 mg tid orally daily

SUMMARY:
R(+)pramipexole is administered in escalating doses to patients with early ALS. Plasma and spinal fluid levels of R(+)PPX are monitored, in addition to biochemical markers of oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* definite ALS no prior exposure to R(+)PPX

Exclusion Criteria:

* ALSFRS at baseline <40 FVC at baseline <70%

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
decline in ALSFRS score | 6 months

SECONDARY OUTCOMES:
plasma PPX levels | 6 months
CSF PPX levels | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ted M Burns, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Result] Wang H, Larriviere KS, Keller KE, Ware KA, Burns TM, Conaway MA, Lacomis D, Pattee GL, Phillips LH 2nd, Solenski NJ, Zivkovic SA, Bennett JP Jr. R+ pramipexole as a mitochondrially focused neuroprotectant: initial early phase studies in ALS. Amyotroph Lateral Scler. 2008 Feb;9(1):50-8. doi: 10.1080/17482960701791234. PMID 18270879